CLINICAL TRIAL: NCT05014321
Title: Evaluation of the Tolerance and the Mode of Administration of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots
Brief Title: Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots PROOF OF CONCEPT
Acronym: CRYO-EC4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry); INNOVSOLUTION (Unknown); CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CRYO-N° 21D588A0001
Record Dates: First submitted 2021-07-12; First posted 2021-08-20 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Lentigo Solar
Keywords: Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each spot will be treated by a defined prototype / device (always the same prototype / device on the same spot all along the study - one unique prototype/device per spot). The application order of the different device prototypes (810A-v1), (810B-v1), (810C-v1) will be defined by randomization except for CNV Body that will always be applied last.
  Each prototype will be identified by a 3 characters internal code (00-x) corresponding to the treated spot with "00" corresponding to the subject number from 01 to 12 and "x" corresponding to the selected spot from A to D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EC16 medical device (CE marked) — Application on brown spots located on the face (1 treatment during the study).
  Other Names: CNV Body
Device: device prototype (810A-v1) — Application on brown spots located on the face (4 treatments during the study).
Device: device prototype (810B-v1) — Application on brown spots located on the face (4 treatments during the study).
Device: device prototype (810C-v1) — Application on brown spots located on the face (4 treatments during the study).

SUMMARY:
CRYO (N° 21D588A0001) study aims to evaluate the tolerance and adjust the mode of administration of a cyto-selective difluoroethane-based cryotherapy in the treatment of brown spots.

The study is a proof of concept on a small panel of subjects and has been designed to be interventional, monocentric, randomized and double blind.

The study will include three device prototypes and a CE marked device (trademark URGO CRYOBEAUTY MAINS-BRAS-JAMBES) used as reference.

DETAILED DESCRIPTION:
Solar lentigo is a harmless patch of darkened skin. It results from exposure to ultraviolet (UV) radiation, which causes local proliferation of melanocytes and accumulation of melanin within the skin cells (keratinocytes). Solar lentigos or lentigines are very common, especially in people over the age of 40 years.

CRYONOVE PHARMA develops and manufactures cryotherapy-based devices to improve skin appearance and treat lentigo spot. The mode of action of CRYONOVE devices consists to "provoke a selective cell death (melanocyte & melanosome) by thermic shock induced by a rapid decrease in skin temperature via the diffusion of difluoroethane gas to the skin".

In this proof of concept study, the sponsor aims to assess the tolerance and the admininistration mode of cryogenic spray which could be used for lentigo treatment on the face.

The study is exploratory, interventional, monocentric, randomized and double blind.

Three prototypes of devices for face are compared to a CE marking device (trademark URGO CRYOBEAUTY MAINS-BRAS-JAMBES) used as reference.

Twelve subjects with at least 4 spots on face are expected to be included, in order to evaluate a minimum of 48 brown spots. Volunteers are treated at T0 only with the reference device and at T0, T2, T4, T6 weeks with the prototype devices. The patient follow-up include 10 visits from D0 to D56.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* Ages 30 to 75.
* Phototype II et III according to Fitzpatrick scale
* Featuring brown spots (solar lentigos) on the face ≥ 3 mm to ≤ 6 mm in diameter (at least 4 spots per subject).
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his ability to participate in the study.
* Having given written consent for participation in the study.
* No suspicion of carcinoma after investigation by a Dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, manicures, facials, UV ...) in the month before the start of the study, at the level of the face.
* Having applied a depraving product in the month prior to the start of the study, at the level of the face.
* Having performed cosmetic treatments in a dermatologist (laser, IPL, peeling, creams, cryotherapy ...), at the level of the face in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write Ukrainian language.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman, who does not use effective methods of contraception.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
TOLERABILITY : Post-treatment pain assessement | Day 0 (Time1 defined as 15 minutes post-treatment)
  The pain of the treatment will be assessed by the VAS (Visual Analogue Scale). Pain intensity is measured in millimeters by the distance from the position of the mark to the "no pain" extremity.
  Based on the distribution of pain VAS scores in postoperative patients, the following bounds were recommended for the assessment of this scale: no pain (0-4mm), mild pain (5-44mm), moderate pain (45-74 mm) and severe pain (75- 100 mm).
  The expected outcomes are pain score < 44 mm (mild pain) for CNV Body and score < 4 mm (no pain) for each prototype.
TOLERABILITY : Appearance of edemas, blisters, bubbles or scars. | Day 56
  Clinical evaluation of treated lentigo spot will be performed by a Dermatologist by scoring with standardized position and lighting.
  The evaluation will be performed visualy on the selected lentigo spots and surrounded spotless skin area around the spot skin.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
  The expected score is < 1.
PERFORMANCE : Skin color evaluation | Day 56
  Clinical evaluation of each treated lentigo spot and spotless area (one on face and far from a lentigo spot) will be performed in blinded conditions by a trained assessor by scoring using L'OREAL ColorChart* in standardized position and lighting.
  The score delta between Day 56 post treatment and D0 pre-treatment will be calculated.
  The expected results is a score delta (D56-D0) < -1 for lighteness of lentigo spot.
  *Jean de Rigal, Marie-Laurence Abella, Franck Giron, Laurence Caisey, Marc André Lefebvre - Development and validation of a new Skin Color Chart® - Skin Research1 Technology, January 2007.

SECONDARY OUTCOMES:
TOLERABILITY : Hyperpigmentation | Day 0/Time 0 to Day 56
  Clinical evaluation of hyperpigmentation on each selected and treated lentigo spot will be performed by a Dermatologist by scoring with standardized position and lighting.
  The evaluation will be performed visualy on the selected lentigo spots. A scale in 6 points (0 to 5) will be used : 0=Clear of hyperpigmentation, 1= Almost clear of hyperpigmentation, 2=mild, but noticeable hyperpigmentation, 3=moderate hyperpigmentation (medium brown in quality), 4=severe hyperpigmentation (dark brown in quality), 5= very severe hyperpigmentation (very dark brown, almost black in quality).
  The expected outcomes are Score ≤ 3 (moderate hyperpigmentation, medium brown in quality) for CNV Body and Score ≤ 2 (mild, but noticeable hyperpigmentation) for each prototype.
TOLERABILITY : Hypopigmentation | Day 0/Time 0 to Day 56
  Clinical evaluation of hyperpigmentation on each selected and treated lentigo spot will be performed by a Dermatologist by scoring with standardized position and lighting.
  The evaluation will be performed visualy on the selected lentigo spots. A scale in 5 points (0 to 4) will be used: 0=no hypopigmented lesion, 1= very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin, 2= slight area of hypopigmentation of small size and slightly fairer than the surrounding skin, 3= moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin, 4= severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
  The expected outcomes are Score ≤ 3 (area of hypopigmentation of moderate size and much fairer than the surrounding skin) for the CNV body device and Score ≤ 2 (slight area of hypopigmentation of small size and slightly fairer than the surrounding skin) for each prototype.
TOLERABILITY : Erythema | Day 0/Time 0 to Day 56
  Clinical evaluation of treated lentigo spot will be performed by a Dermatologist by scoring with standardized position and lighting.
  The evaluation will be performed visualy on the selected lentigo spots and surrounded spotless skin area around the spot skin.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
  The expected score is ≤ 3 (moderate) for the CNV body device and score ≤ 2 (mild) for each prototype device.
TOLERABILITY : Skin sensation | Day 0/Time 0 to Day 56
  The dermatologist will collect functional signs by asking the subjects about tightness, stinging, itching, warm or burning sensation.
  The evaluation will be performed visualy regarding the selected lentigo spots and surrounded spotless skin area around the spot skin.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
  The expected score is ≤ 3 (moderate) for the CNV body device and score ≤ 2 (mild) for each prototype device.
PERFORMANCE: Standardized photographs by C-Cube® acquisition | Day 56
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE).
  The capture will be taken on the previously selected lentigo (and spotless surrounding each spot in the same acquisition) and a spotless area (one on face (same as clinical evaluation) and far from a lentigo spot). Acquisition will be performed at Day0/time 0 (before treatment) and at each visit.
  The expected outcomes at day 56 are a score delta (D56-D0) > 2,5 for ITA of lentigo spot for the CNV Body device and a score delta (D56-D0) > 2 for ITA of lentigo spot for the prototype devices.
EFFICACY: Self-assessment of the subject | From Day 2 to Day 42
  Data will be completed by a questionnaire elaborated by the sponsor and filled in by subjects.
  It allowed obtaining the subjective appraisal of subject on tested laser act using the following 5-point scale: agree; quite agree; neither agree, nor disagree; quite disagree; disagree.
  The items are the following:
  * The spot seems clearer.
  * The size of the spot seems reduced.
  * The spot seems less visible.
  The expected results are subject appraisal at day 42 "agree" on the 3 parameters a for the CNV Body device and "agree" or "quite agree" on the 3 parameters for the prototype devices.
TOLERABILITY: other expected events | Day 0/Time 0 to Day 56
  Clinical evaluation of treated lentigo spot will be performed by a Dermatologist regarding dryness, desquamation, fissures, cracks, roughness or crust. The evaluation will be done visualy by scoring on the selected lentigo spots and surrounded spotless skin area around the spot skin, with standardized position and lighting.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
  The expected score is ≤ 3 (moderate) for the CNV body device and score ≤ 2 (mild) for each prototype device.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Didenko, MD, Principal Investigator — VIDNOVLENNYA invetigation site
Locations (1):
- Vidnovlennya, Zhytomyr, Ukraine

IPD SHARING:
Plan to Share IPD: No